CLINICAL TRIAL: NCT02392650
Title: Microbiome And Multi'Omics In Preterm Birth: The Bacteria And Birth Study (BaBs)
Brief Title: Microbiome And Multi'Omics In Preterm Birth: The Bacteria And Birth Study
Acronym: BaBs
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Baylor College of Medicine (Other)
Collaborators: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Principal Investigator, Kjersti Aagaard, Associate Professor, Maternal-Fetal Medicine and Vice Chair for Research at Baylor College of Medicine, Baylor College of Medicine
Other Study IDs: H-34056
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Samples with DNA, RNA and metabolites
Oversight: Data Monitoring Committee: No

SUMMARY:
Hominids and hominins serve as remarkable hosts to microbes, and we have co-evolved over the past 4.5 million years as highly plethoric communities. Human-associated microorganisms (the "microbiome") are present in numbers exceeding the quantities of human cells by at least 10-fold beginning in the neonatal period. The collective genome (the "metagenome") exceeds our human genome in terms of gene content by more than 150-fold. With respect to microbiota and preterm birth, it has generally assumed that the majority of intrauterine infections originate in the lower genital tract, with microbiota ascending into the otherwise sterile intrauterine environment to infect the placenta (preterm birth), fetal membranes (chorioamnionitis), umbilical cord (funisitis), and the fetus (sepsis). However, we and others have recently demonstrated that the vaginal and gut microbiome communities are distinctly structured in pregnancy, and the placenta is in fact not sterile, but rather harbors a low-abundance microbiome which is likely acquired through hematogenous transmission of the oral microbiome.

Based on our prior studies and preliminary data, our central hypothesis is that a distinct and largely commensal resident microbiome in pregnancy renders risk for preterm birth. By utilizing our state-of-the-science technology and analysis tools in a longitudinal case-cohort of preterm birth subjects, we will be able to transform "discovery based" metagenomics and multi'omics science into readily translatable mechanistic studies at a previously unparalleled level.

DETAILED DESCRIPTION:
Specific Aim 1. Longitudinal maternal (vaginal, oral, skin, gut), fetal (oral, skin, gut) and placental (basal plate and parenchyma) 16S-based metagenomic profiling with inferred metagenomics will reveal distinct microbial communities in association with preterm birth. Methods: We will enroll 526 at-risk gravidae to yield an approximated 135 preterm births with 401 at-risk term controls. Starting in the first/early second trimester, we will sample multiple body sites (vagina, oral, stool, placenta) at multiple time points (antenatal through delivery), isolate microbial DNA, and perform 16S-based determination of niche-specific microbial communities found in association with preterm birth. With our case-cohort longitudinal design, we will be able to apply our well-developed supervised learning approaches to reveal which taxa contribute to risk of preterm birth, and at what body sites and gestational ages they are predictive of preterm birth.

Specific Aim 2. Whole-genome shotgun (WGS) metagenomics from selected subjects and body sites will enable species identification, generation of microbial gene catalogues, and metabolic reconstructions to determine the structure, function and diversity of the preterm birth microbiome. Methods: To probe metabolic functionality and describe pathogen-related mechanisms, we will analyze changes in total gene content using shotgun metagenomics on a subset of samples. We will build on our functional computational pipelines to fully characterize targeted subjects' metagenomic signatures.

Specific Aim 3. Integrated host genomics, metatranscriptomics and metabonomics data will reveal molecular mechanisms and networks underlying preterm birth in a limited subset of samples. Methods: We will interrogate and integrate our concomitantly acquired clinical metadata, microbial and host gene expression data (RNA-Seq metatranscriptomics), and metabonomics profiling with advanced computational and biostatistical approaches. We will be guided in our choice of subjects by our data from Aims 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Gravidae at risk for preterm birth, defined as: History of prior spontaneous preterm birth at 16w0d-36w6d gestational age confirmed by review of medical records. If efforts to retrieve medical records are unsuccessful, eligibility will depend upon the events surrounding the prior birth and birthweight under 2 kg; Documented shortened cervix <2.5 cm by transvaginal ultrasound performed by experienced sonographer at <24 weeks gestational age; Documented and culture-proven complicated lower or upper urinary tract infection defined as a urinary tract infection requiring hospitalization (e.g., pyelonephritis); Documented periodontal disease, treated or untreated; Documented recurrent lower genital infection; Smoking or other chemical dependency that would convey an increased risk of preterm birth; Other clinical concern for high risk of preterm birth (and cleared by PI Dr. Aagaard at BCM or Dr. Saade at UTMB)
* Enrollment at less than or equal to 20 weeks gestation by best obstetrical estimate
* Able to speak English or work with an interpreter
* Cognitively aware enough to be able to participate in the study
* Gravidae with viable pregnancy >10 weeks gestational age
* Willingness to consent to all required aspects of protocol - There will be additional non-required aspects that we will recruit 20% of subjects to participate in. These will be voluntary opt-in aspects
* 16 years of age or older

Exclusion Criteria:

* Multifetal gestation at any time during the pregnancy
* Known HIV or Hepatitis C infection
* Known immunosuppressive disease
* Use of any of the following drugs within the last 6 months; Cytokines; Methotrexate or immunosuppressive cytotoxic agents
* History of cancer except for squamous or basal cell carcinomas of the skin or thyroid cancer that have been managed and fully treated.
* Major surgery of the GI tract (including gastric bypass), with the exception of cholecystectomy and appendectomy in the past five years. Any major bowel resection at any time. If conditions arise that require such surgeries during participation in the study, subjects will not be excluded after enrollment. If patient develops need for such surgery after enrollment, they will not be excluded.
* Documented chronic GI disorders, (e.g., Crohn's diseae)
* Chronic conditions with GI symptoms, (e.g. cystic fibrosis)
* Autism spectrum disorder or significant developmental delay, psychosis, major depressive disorder, or a history of bipolar disorder if there is concern about ability to consent
* Treatment for or suspicion of ever having had toxic shock syndrome.
* Fatal fetal anomaly. Will exclude after enrollment if not previously identified

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women who are currently pregnant who are at high risk for preterm birth; Pregnant with one baby (not twins or triplets) and who attend regular prenatal visits. They will spend an extra 20 minutes at 5-6 priority scheduled visits to obtain study samples and complete questionnaires, with the last visit occurring around 6 weeks after delivery.
Sampling Method: Non-Probability Sample
Enrollment: 526 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Characterization of Maternal-Fetal microbiome | Conception to 4-6 weeks postpartum
  Longitudinally characterize the maternal, placental, and infant microbiome in a cohort at risk of preterm birth. Not all the women will ultimately deliver preterm; we we will be able to see if there are microbiome changes associated with preterm birth.
Association of maternal microbiome (gut, oral, vaginal, placenta) with preterm birth | Conception to 4-6 weeks postpartum
  Longitudinally characterize the maternal, placental, and infant microbiome in a cohort at risk of preterm birth. Not all the women will ultimately deliver preterm; we we will be able to see if there are microbiome changes associated with preterm birth.

SECONDARY OUTCOMES:
Rate of Preterm Birth | Conception to date of date of delivery, <37 weeks
  Measure rate of preterm birth <37 and <34 weeks gestation, as defined by best obstetrical estimate of last menstrual period consistent with <24 week sonogram, OR <24 week sonogram with unknown last menstrual period, OR skilled examination and <24 week sonogram
Rate of Term Birth | Conception to date of date of delivery
  Measure rate of term birth, as defined by best obstetrical estimate of last menstrual period consistent with <24 week sonogram, OR <24 week sonogram with unknown last menstrual period, OR skilled examination and <24 week sonogram

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti Aagaard, MD/PhD, Principal Investigator — Associate Professor / Vice Chair for Research
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States